CLINICAL TRIAL: NCT04132882
Title: A Compassionate Use Program to Provide Access to Sodium Thiosulfate for the Protection From Cisplatin-Induced Hearing Loss in Children Who Had Standard-risk Hepatoblastoma
Brief Title: A Compassionate Use Program to Provide Access to Sodium Thiosulfate
Status: Available | Type: Expanded Access
Sponsor: TRPHARM (Industry)
Collaborators: Fennec Pharma (Unknown)
Responsible Party: Sponsor
Other Study IDs: TRP-STS-001
Record Dates: First submitted 2019-10-16; First posted 2019-10-21 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Cisplatin-Induced Hearing Loss in Children Who Had Standard-risk Hepatoblastoma
Keywords: Cisplatin; Hearing Loss; Hepatoblastoma
MeSH Terms: conditions — Hearing Loss; Hepatoblastoma | interventions — sodium thiosulfate

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Sodium Thiosulfate (STS)

SUMMARY:
This is a CUP which is designed to provide treatment access of STS to pediatric patients for the protection from Cisplatin-Induced Hearing Loss in children who had standard-risk hepatoblastoma.

Approximately 10 patients will be treated as part of this program as specified below:

Sodium Thiosulfate vials i.v. 80 mg/mL.

This Compassionate Use Program for STS will consist of 2 phases:

Screening:

Patients will only be able to participate in this CUP if they meet the eligibility criteria.

Treatment:

Any clinical assessments, physical examinations, and dosage changes will be determined by the treating physician as per local standard medical practice.

All serious adverse events (SAEs) will be reported. All related non-serious adverse events (AEs) will be reported where "related" means any event where a causal relationship between STS and the event is at least, a reasonable possibility. All non-serious AEs leading to dose modification or discontinuation will be reported. Pregnancies, outcomes of pregnancies, and exposure through breastfeeding will also be reported.

ELIGIBILITY:
Inclusion Criteria:

I-1. Children older than 1 month and younger than 18 years of age who had standard-risk hepatoblastoma that had not been treated previously with STS and receive cisplatin.

I-2. A written informed consent was provided from all the patients and/or parents or legal guardians of children.

Exclusion Criteria:

E-1. Any previous participation in an STS clinical trial. E-2. Participation in another clinical study with an investigational product during the most recent chemotherapy course.

E-3. Patients with a known hypersensitivity to STS or any of the excipients of the product.

E-4. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) or major surgery within 3 weeks prior to STS treatment.

E-5. Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) CTCAE grade 2) caused by previous cancer therapy, excluding alopecia.

E-6. Breast feeding or pregnant women.

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University School of Medicine, Ankara, Turkey (Türkiye)